CLINICAL TRIAL: NCT06061432
Title: Endoscopic Reconstruction of the Gastrointestinal Tract After Surgical Resection Procedures Within the Large Intestine (Hartmann's Procedure- Modification of the Method Facilitating the Restoration of Gastrointestinal Continuity)
Brief Title: Endoscopic Ultrasound- Guided Hartmann Reversal Procedure
Acronym: EndoHARP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nicolaus Copernicus University (Other)
Collaborators: Medical University of Łódź (Other)
Responsible Party: Principal Investigator, Mateusz Jagielski, Professor, Nicolaus Copernicus University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DGGOS/MJ/1/2023
Record Dates: First submitted 2023-09-12; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Colorectal Neoplasms; Diverticular Diseases; Inflammatory Bowel Diseases
Keywords: colorectal surgery; endotherapy; anastomosis; endoscopic ultrasound; gastrointestinal continuity; Hartmann procedure
MeSH Terms: conditions — Colorectal Neoplasms; Diverticular Diseases; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endoscopic Ultrasound- Guided Hartmann Reversal Procedure (Experimental): Participants after Hartmann procedure, who were qualified and underwent Endoscopic Ultrasound- Guided Hartmann Reversal Procedure.
  Interventions: Procedure: Endoscopic restoration of gastrointestinal continuity after Hartmann procedure

INTERVENTIONS:
Procedure: Endoscopic restoration of gastrointestinal continuity after Hartmann procedure — EndoHARP is a new technique proposed to restore gastrointestinal continuity after the Hartmann's procedure. For EndoHARP, a fixed loop of the large intestine will be identified on endosonography after an echoendoscope is inserted into the rectal stump under endoscopic guidance. Then, using the set for inserting self-expandable metal transmural endoprosthesis (20 mm in diameter and 10 mm in length) with electrocautery (as in endoscopic gastroenterostomy), EUS-guided anastomosis of the rectal stump to the large intestine loop will be performed, allowing the natural passage of intestinal contents through the endoscopic anastomosis, restoring gastrointestinal continuity. The aim of leaving the self-expandable transmural endoprosthesis in the anastomosis is not only to maintain the patency of the intestinal anastomosis of at least 20 mm in diameter, but also to diminish the risk of endoscopic intestinal anastomotic leak by completely covering the prosthesis with a polymer layer.

SUMMARY:
The goal of this clinical trial is to learn about clinical usefulness endoscopic gastrointestinal anastomoses to restore the gastrointestinal continuity in patients with permanent colostomy after Hartmann procedure.

The main questions it aims to answer are:

* is the endoscopic restore the gastrointestinal continuity procedure effective?
* is this endoscopic procedure safe?

DETAILED DESCRIPTION:
Large intestinal resection is performed for both elective and acute reasons. The choice of surgical technique is determined not only by the oncological treatment outcome, but also by the patient's quality of life after surgery. Intestinal anastomosis is associated with the risk of leakage, which is one of the most serious complications of colorectal surgery. In the event of this complication, the most common treatments are relaparotomy/relaparoscopy and disconnection of the anastomosis with stoma formation. The patient's condition is most often critical, and the mortality associated with this complication ranges from 1.3 to 27% depending on the patient's age. In addition, dehiscence of the intestinal anastomosis during oncological surgery is an independent factor that increases the risk of local recurrence and shortens disease-related survival. In contrast, avoiding primary anastomosis and performing Hartmann's surgery (resection with the formation of an end colostomy) is safer for the patient as there is no risk of anastomotic leak. However, this procedure is not ideal. The patient undergoes an end colostomy, which is often difficult for the patient to accept, especially during the initial period. Restoration of gastrointestinal continuity is possible a few months after primary surgery. In colorectal cancer, it can be treated only after the completion of adjuvant chemotherapy, which significantly prolongs this process. Stoma closure has never been attempted in many patients because of the risks associated with another major surgery. Therefore, it is not surprising that there is a trend towards performing primary anastomosis. In experienced centers, the risk of anastomotic dehiscence is at an acceptable level of less than 5% for elective surgeries. In contrast, the percentage is higher for acute surgeries, accounting for up to 20% of emergency indications, especially in centers inexperienced in colorectal surgery. Gastrointestinal obstruction, which is most often associated with colorectal tumors, leads to dilatation of the proximal segment of the large intestine (above the tumor) with wall thickening. Disproportion in diameter, edema, thickening of the intestinal wall, and serious conditions with accompanying malnutrition significantly increased the risk of anastomotic leak in this group of patients. Currently, due to advances in pharmacological treatment and interventional radiology (percutaneous abscess drainage), surgical treatment involving segmental intestinal resection is reserved for patients with diffuse peritonitis. In this group of patients, resection with a primary anastomosis is associated with a very high risk of anastomotic failure, and Hartmann's resection remains the safest option.

Previous methods for restoring gastrointestinal continuity after Hartmann's procedure required extensive surgery. The first stage of surgery involves the dissection of adhesions after the previous resection. It is usually the most technically difficult stage of the procedure because of the emergency nature of the primary surgery (obstruction/peritonitis). Once the intestinal adhesions are removed, the colostomy is dissected from the wall, and the descending and sigmoid colons are mobilized. This is most often associated with the need to release splenic flexure. The next step is to identify and mobilize the rectal stump. This is necessary for a safe intestinal anastomosis, which is most often performed using a circular stapler. If a long rectal stump remains after the primary surgery, insertion of the stapler into its terminal segment is sometimes difficult and involves dissection and cutting of the pelvic peritoneum. Restoring gastrointestinal continuity after Hartmann's surgery is technically difficult and carries a high risk of intra- and perioperative complications, with the most common being small/large intestinal injury during adhesion dissection, intraoperative bleeding, ureteral/bladder injury, and splenic injury (most often, the splenic flexure needs to be released). No technical possibility of reconstruction is common (displacement of the rectal stump deep inside the pelvis and shortening of the mesentery of the left half of the colon). The risk of complications related to the restoration of gastrointestinal continuity after Hartmann's surgery is 30-60%; thus, a significant number of patients do not consent to this procedure.

The endoHARP procedure proposed in this article allows easier restoration of gastrointestinal continuity owing to the combination of classic colorectal surgical techniques with endosonography techniques. The technical details of the procedure are described later in this article. To ensure the feasibility of the endoHARP procedure, it is necessary to slightly modify the primary resection procedure using Hartmann's method. After the resection stage, which does not differ from the original surgery, the remaining parts of the sigmoid and descending colon should be mobilized at the promontorium level. This allows fixation of the closed rectal stump. Side-to-end anastomosis of the intestine to the rectal stump was performed using four 3-0 absorbable sutures. The end of the sigmoid colon is typically brought out into the left middle abdomen. However, this procedure may not be feasible for all patients. It is not possible to use this modification in most cases involving a short segment of the remaining left half of the colon, those with inflammatory infiltration within the mesentery, or those requiring anterior rectal resection (low-sigmoid tumors). However, this modification is technically feasible in a considerable number of patients undergoing Hartmann's procedure.

The steps of the modified Hartmann's sigmoid resection procedure are summarized below.

1. Resection of the sigmoid colon performed as in the original method
2. Mobilization of the remaining part of the sigmoid and descending colon
3. Possible mobilization of the splenic flexure
4. Fixation of the descending and sigmoid colon to the rectal stump with four 3-0 serous sutures

Endoscopic ultrasound (EUS)-guided restoration of gastrointestinal continuity At least 12 weeks (ranging from 3 to 6 months) should elapse between the formation of the colostomy and its closure (i.e., restoration of gastrointestinal continuity). The classic method for the restoration of gastrointestinal continuity involves opening the abdominal cavity, dissection of the intestinal stump and stoma and its closure, enteroenteric anastomosis with manual or mechanical sutures, and closure of the abdominal cavity. However, during the restoration of gastrointestinal continuity after opening the abdominal cavity, the surgeon usually finds numerous adhesions from the previous surgery, which technically impedes the procedure and requires careful dissection to avoid iatrogenic intestinal perforation. In some cases, anatomical conditions encountered after opening the abdominal cavity prevent surgery. The patient is then destined to have a permanent stoma because the restoration of gastrointestinal continuity is technically impossible. In addition, surgical procedures to restore gastrointestinal continuity are associated with the risk of enteroenteric anastomotic leakage.

Recent developments in interventional endoscopy of the gastrointestinal tract and the therapeutic use of EUS have enabled endoscopic gastrointestinal anastomoses using transmural self-expandable prostheses to restore gastrointestinal continuity in patients with high gastrointestinal obstruction. During EUS-guided gastroenterostomy, the gastric lumen is anastomosed to the small intestinal lumen (gastrointestinal anastomosis). Endoscopic anastomosis of the stomach to the small intestine in patients with high gastrointestinal obstruction is performed by inserting a self-expandable metal transmural endoprosthesis (20 mm in diameter and 10 mm in length) using electrocautery under endoscopic, fluoroscopic, and endosonography guidance. A similar approach will be used in our EndoHARP technique to restore gastrointestinal continuity after the Hartmann's procedure. For EndoHARP, a fixed loop of the large intestine will be identified on endosonography after an echoendoscope is inserted into the rectal stump under endoscopic guidance. In addition, a contrast agent administered through colostomy will fill the intestinal loop which will be visible on both EUS and fluoroscopy, improving visibility during endoscopic surgery. Then, using the set for inserting self-expandable metal transmural endoprosthesis (20 mm in diameter and 10 mm in length) with electrocautery (as in endoscopic gastroenterostomy), EUS-guided anastomosis of the rectal stump to the large intestine loop will be performed, allowing the natural passage of intestinal contents through the endoscopic anastomosis, restoring gastrointestinal continuity. The aim of leaving the self-expandable transmural endoprosthesis in the anastomosis is not only to maintain the patency of the intestinal anastomosis of at least 20 mm in diameter, but also to diminish the risk of endoscopic intestinal anastomotic leak by completely covering the prosthesis with a polymer layer.

After endoscopic surgery, the patients will undergo a gastrointestinal passage examination with a contrast agent for four weeks. If the patency of the endoscopic enterorectal anastomosis is confirmed radiologically, the patient will be eligible for colostomy closure in a traditional surgical procedure (i.e., cutting and closing the colostomy with a linear stapler, returning it to the abdominal cavity without the need for intestinal dissection, removal of peritoneal adhesions, and most importantly, for intestinal anastomosis). Thus, the risks of intestinal anastomotic leakage and iatrogenic intestinal perforation during dissection are avoided, thereby increasing the safety of the procedure. Then, the skin area after colostomy will be closed in layers. The metal endoprosthesis will be simultaneously removed from the enterorectal anastomosis during the surgical closure of the colostomy. At this point, the interventional treatment is completed, and gastrointestinal continuity is permanently restored.

The patient will be followed up periodically in the Surgical Clinic every 3 months for the first 12 months after surgery and every 6 months for the next 4 years. Follow-up endoscopic examinations of the lower gastrointestinal tract with evaluation of enterorectal anastomosis will be scheduled every 3-6-12 months, and then every 3 years for the next 9 years.

Number of participants necessary to demonstrate an effect is 100.

The stages of EUS-guided restoration of gastrointestinal continuity are summarized below.

THE FIRST STAGE of endoscopic restoration of gastrointestinal continuity

1. Administration of a contrast agent through the stoma to the intestinal loop
2. Insertion of the echoendoscope into the rectal/colon stump and identification of fixed and contrast-filled large/small intestinal loops on EUS
3. Performance of EUS-guided enterorectal/enteroenteric anastomosis using a set for inserting a self-expandable metal transmural endoprosthesis with electrocautery

   1. performance of a transmural/transrectal puncture using electrocautery
   2. expansion of the transmural endoprosthesis through the puncture site
   3. contrast administration through anastomosis to confirm the tightness of enterorectal/enteroenteric anastomosis
   4. Extend the transmural endoprosthesis lumen with a high-pressure balloon up to 20 mm in diameter.

THE SECOND STAGE (after four weeks) of endoscopic restoration of gastrointestinal continuity

One surgical team

1. Circular incision around the stoma
2. Closure of colostomy with a linear stapler
3. Return of the closed intestinal loop into the abdominal cavity
4. Skin closure

Simultaneously - second surgical team (endoscopic)

1. Insertion of the endoscope into the rectum
2. Seizure of the transmural endoprosthesis with endoscopic forceps
3. Removal of the endoprosthesis
4. Endoscopic and fluoroscopic follow-up of endoscopic intestinal anastomosis

ELIGIBILITY:
Inclusion Criteria:

* participants of both sexes aged above 18 years
* participants, who provided informed consent for such treatment
* eligibility for Hartmann's procedure according to current medical knowledge based on evidence-based medicine.

Exclusion Criteria:

* pregnancy, breastfeeding, or intention to become pregnant during the study
* contraindications to electrosurgical instruments
* allergy to any of the materials used in the study
* participants with advanced cancer in the metastatic stage
* participants ineligible for restoration of gastrointestinal continuity
* participants ineligible for surgery
* participants ineligible for general anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of efficacy of endoscopic gastrointestinal anastomoses using transmural self-expandable prostheses to restore the gastrointestinal continuity in patients after Hartmann procedure (Endo-HARP) | 12 months
  Evaluation of efficacy based on patency of endoscopic entero-rectal anastomosis confirmed radiologically and endoscopically.
  Unit of Measure: the number of participants with patency of endoscopic entero-rectal anastomosis compared to the total number of participants, who underwent endoscopic gastrointestinal anastomoses using transmural self-expandable prostheses to restore the gastrointestinal continuity in patients after Hartmann procedure (Endo-HARP)
Rate of complications during endoscopic gastrointestinal anastomoses using transmural self-expandable prostheses to restore the gastrointestinal continuity in patients after Hartmann procedure (Endo-HARP) | 12 months
  Evaluation of all complications in patients with endoscopic gastrointestinal anastomoses (Endo-HARP).
  Unit of Measure: the number of participants with complications compared to the total number of participants, who underwent endoscopic gastrointestinal anastomoses using transmural self-expandable prostheses to restore the gastrointestinal continuity in patients after Hartmann procedure (Endo-HARP).

SECONDARY OUTCOMES:
Rate of early complications during endoscopic gastrointestinal anastomoses using transmural self-expandable prostheses to restore the gastrointestinal continuity in patients after Hartmann procedure (Endo-HARP) | 30 days
  Evaluation of early complications within thirty days from onset of endoscopic gastrointestinal anastomoses (Endo-HARP) procedure.
  Unit of Measure: the number of participants with early complications compared to the total number of participants, who underwent endoscopic gastrointestinal anastomoses using transmural self-expandable prostheses to restore the gastrointestinal continuity in patients after Hartmann procedure (Endo-HARP).
Rate of late complications during endoscopic gastrointestinal anastomoses using transmural self-expandable prostheses to restore the gastrointestinal continuity in patients after Hartmann procedure (Endo-HARP) | 12 months
  Evaluation of late complications after thirty days from onset of endoscopic gastrointestinal anastomoses (Endo-HARP) procedure.
  Unit of Measure: the number of participants with late complications compared to the total number of participants, who underwent endoscopic gastrointestinal anastomoses using transmural self-expandable prostheses to restore the gastrointestinal continuity in patients after Hartmann procedure (Endo-HARP).
Rate of technical success of endoscopic gastrointestinal anastomoses using transmural self-expandable prostheses to restore the gastrointestinal continuity in patients after Hartmann procedure (Endo-HARP) | duration of procedure
  Assessment of correct conduct of endoscopic gastrointestinal anastomoses using transmural self-expandable prostheses to restore the gastrointestinal continuity in patients after Hartmann procedure (Endo-HARP) according to study protocol.
  Unit of Measure: the number of participants with technical success to the total number of participants, who underwent endoscopic gastrointestinal anastomoses using transmural self-expandable prostheses to restore the gastrointestinal continuity in patients after Hartmann procedure (Endo-HARP).
Rate of clinical success of endoscopic gastrointestinal anastomoses using transmural self-expandable prostheses to restore the gastrointestinal continuity in patients after Hartmann procedure (Endo-HARP) | 12 months
  Assessment of clinical results of endoscopic gastrointestinal anastomoses using transmural self-expandable prostheses to restore the gastrointestinal continuity in patients after Hartmann procedure (Endo-HARP).
  Unit of Measure: the number of participants with clinical success to the total number of participants, who underwent endoscopic gastrointestinal anastomoses using transmural self-expandable prostheses to restore the gastrointestinal continuity in patients after Hartmann procedure (Endo-HARP).

CONTACTS AND LOCATIONS:
Overall Officials: Mateusz Jagielski, Prof., Principal Investigator — Department of General, Gastroenterological and Oncological Surgery, Collegium Medicum, Nicolaus Copernicus University in Toruń, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zaimi I, Sparreboom CL, Lingsma HF, Doornebosch PG, Menon AG, Kleinrensink GJ, Jeekel J, Wouters MWJM, Lange JF; Dutch ColoRectal Audit Group. The effect of age on anastomotic leakage in colorectal cancer surgery: A population-based study. J Surg Oncol. 2018 Jul;118(1):113-120. doi: 10.1002/jso.25108. Epub 2018 Jun 7. PMID 29878360
- [Background] Bakker FC, Hoitsma HF, Den Otter G. The Hartmann procedure. Br J Surg. 1982 Oct;69(10):580-2. doi: 10.1002/bjs.1800691007. PMID 7127036
- [Background] Hallam S, Mothe BS, Tirumulaju R. Hartmann's procedure, reversal and rate of stoma-free survival. Ann R Coll Surg Engl. 2018 Apr;100(4):301-307. doi: 10.1308/rcsann.2018.0006. Epub 2018 Feb 27. PMID 29484943
- [Background] Mirnezami A, Mirnezami R, Chandrakumaran K, Sasapu K, Sagar P, Finan P. Increased local recurrence and reduced survival from colorectal cancer following anastomotic leak: systematic review and meta-analysis. Ann Surg. 2011 May;253(5):890-9. doi: 10.1097/SLA.0b013e3182128929. PMID 21394013
- [Background] Zarnescu EC, Zarnescu NO, Costea R. Updates of Risk Factors for Anastomotic Leakage after Colorectal Surgery. Diagnostics (Basel). 2021 Dec 17;11(12):2382. doi: 10.3390/diagnostics11122382. PMID 34943616
- [Background] Tsalikidis C, Mitsala A, Mentonis VI, Romanidis K, Pappas-Gogos G, Tsaroucha AK, Pitiakoudis M. Predictive Factors for Anastomotic Leakage Following Colorectal Cancer Surgery: Where Are We and Where Are We Going? Curr Oncol. 2023 Mar 7;30(3):3111-3137. doi: 10.3390/curroncol30030236. PMID 36975449
- [Background] Jaruvongvanich V, Mahmoud T, Abu Dayyeh BK, Chandrasekhara V, Law R, Storm AC, Levy MJ, Vargas EJ, Marya NB, Abboud DM, Ghazi R, Matar R, Rapaka B, Buttar N, Truty MJ, Aerts M, Messaoudi N, Kunda R. Endoscopic ultrasound-guided gastroenterostomy for the management of gastric outlet obstruction: A large comparative study with long-term follow-up. Endosc Int Open. 2023 Jan 13;11(1):E60-E66. doi: 10.1055/a-1976-2279. eCollection 2023 Jan. PMID 36644538
- [Background] Mintziras I, Miligkos M, Wachter S, Manoharan J, Bartsch DK. Palliative surgical bypass is superior to palliative endoscopic stenting in patients with malignant gastric outlet obstruction: systematic review and meta-analysis. Surg Endosc. 2019 Oct;33(10):3153-3164. doi: 10.1007/s00464-019-06955-z. Epub 2019 Jul 22. PMID 31332564
- [Background] Reali C, Landerholm K, George B, Jones O. Hartmann's Reversal: Controversies of a Challenging Operation. Minim Invasive Surg. 2022 Nov 9;2022:7578923. doi: 10.1155/2022/7578923. eCollection 2022. PMID 36406794
- [Background] Mege D, Manceau G, Beyer-Berjot L, Bridoux V, Lakkis Z, Venara A, Voron T, Brunetti F, Sielezneff I, Karoui M; AFC (French Surgical Association) Working Group. Surgical management of obstructive right-sided colon cancer at a national level results of a multicenter study of the French Surgical Association in 776 patients. Eur J Surg Oncol. 2018 Oct;44(10):1522-1531. doi: 10.1016/j.ejso.2018.06.027. Epub 2018 Jul 6. PMID 30041941